CLINICAL TRIAL: NCT01120639
Title: A Phase 1-2 Trial of Temozolomide and Hypofractionated Radiotherapy in Treatment of Supratentorial Glioblastoma Multiforme
Brief Title: Phase 1-2 of Temozolomide and Hypofractionated Radiotherapy in Tx of Supratentorial Glioblastoma Multiform
Acronym: Tx-Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Scott Soltys, Assistant Professor of Radiation Oncology, Stanford University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-17774; SU-04202010-5726 (Other: Stanford University); BRN0012 (Other: OnCore); IRB-17774 (Other: Stanford IRB)
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Glioblastoma; Cancer of Brain and Nervous System; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Neurologic Manifestations | interventions — Temozolomide; Radiosurgery

STUDY DESIGN:
Intervention Model Description: Dose-escalation with 2-level stratification
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stereotactic Radiosurgery (25 Gray x 5 fractions)+Temozolomide (Experimental): Hypofractionated stereotactic radiosurgery with concurrent temozolomide, stratified by Planning Target Volume (PTV) < 60 cm³ vs 60 to 150 cm³.
  Interventions: Drug: Temozolomide; Procedure: Stereotactic Radiosurgery (SRS)
- Stereotactic Radiosurgery (30 Gray x 5 fractions)+Temozolomide (Experimental): Hypofractionated stereotactic radiosurgery with concurrent temozolomide, stratified by Planning Target Volume (PTV) < 60 cm³ vs 60 to 150 cm³.
  Interventions: Drug: Temozolomide; Procedure: Stereotactic Radiosurgery (SRS)
- Stereotactic Radiosurgery (35 Gray x 5 fractions)+Temozolomide (Experimental): Hypofractionated stereotactic radiosurgery with concurrent temozolomide, stratified by Planning Target Volume (PTV) < 60 cm³ vs 60 to 150 cm³.
  Interventions: Drug: Temozolomide; Procedure: Stereotactic Radiosurgery (SRS)
- Stereotactic Radiosurgery (40 Gray x 5 fractions)+Temozolomide (Experimental): Hypofractionated stereotactic radiosurgery with concurrent temozolomide, stratified by Planning Target Volume (PTV) < 60 cm³ vs 60 to 150 cm³.
  Interventions: Drug: Temozolomide; Procedure: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Drug: Temozolomide — 75 mg/m²/day oral, administered concurrently with radiotherapy and as adjuvant therapy.
  Other Names: Temodar; Temodal
Procedure: Stereotactic Radiosurgery (SRS) — Standard of care therapeutic radiotherapy administrated at 25, 30, 35, or 40 Gray (Gy)
  Other Names: Hypofractionated stereotactic radiosurgery (h-SRS); Hypofractionated stereotactic radiotherapy; Cyberknife surgery

SUMMARY:
The purpose of this study is to investigate the safety and effectiveness of a combination treatment for glioblastoma multiforme utilizing radiotherapy plus the FDA-approved chemotherapy drug temozolomide

DETAILED DESCRIPTION:
Primary Objective: To determine the maximum tolerated dose (MTD), based on acute CNS toxicity at 30 days, of hypofractionated radiotherapy given in 5 fractions with temozolomide for the treatment of glioblastoma multiforme.

Secondary Objectives:

1. Assess the short- and long-term adverse effects.
2. Determine the radiographic response rate.
3. Determine the overall survival rate.
4. Assess quality of life during treatment

To determine the maximum tolerated dose (MTD) of hypofractionated (5 fractions) radiotherapy with temozolomide for the treatment of glioblastoma multiforme, patients will be evaluated by a multi-disciplinary team composed of radiation oncologists, neurosurgeons, and neuro-oncologists to assess for their eligibility. Patient's oncologic history, presenting symptoms, physical examination, pathology, and imaging studies will be reviewed. Patients will be evaluated for surgical candidacy and resectability. Patients who are surgical candidates will undergo a surgical resection prior to radiotherapy. Patients whose tumors are unresectable or are not good surgical candidates will undergo a biopsy for tissue diagnosis. Radiation will be delivered in five fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed newly diagnosed glioblastoma multiforme. Diagnosis must be made by surgical biopsy or excision
* The tumor must be supratentorial in location
* The planning target volume (tumor plus margin) must measure ≤ 150 cm^3 in volume
* Age ≥ 18 years
* Life expectancy of at least 12 weeks
* Patient must have adequate organ function to tolerate temozolomide (details in the protocol)

Exclusion Criteria:

* Patients who have previously been treated with brain irradiation to the region that would result in overlap of the radiation fields
* Tumor foci detected below the tentorium
* Multifocal disease or leptomeningeal spread
* Prior allergic reaction to the study drugs involved in this protocol
* Patients with pacemaker will be allowed to undergo CT instead of MRI
* Pediatric patients (age < 18), pregnant women, and nursing patients will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2016-11 (Actual); Study Completion 2020-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gerard Soltys, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Started | 6 | 6 | 6 | 12
Completed | 6 | 6 | 6 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide | Total
Number analyzed (Participants) | 6 | 6 | 6 | 12 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 3 | 5 | 14
  >=65 years | 4 | 2 | 3 | 7 | 16
Age, Continuous [Median (Standard Deviation); unit: Years] | 72 (5.8) | 61.4 (8.3) | 62.8 (10.0) | 67.1 (8.6) | 65.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 4 | 4 | 15
  Male | 2 | 3 | 2 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 12 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicities (DLTs)
Description: The maximum-tolerated dose (MTD) of study treatment (temozolomid plus hypofractionated radiotherapy administered as 5 fractions) is defined as either:
  * The highest radiation dose per protocol, or
  * The radiation dose at which dose-limiting toxicities (DLTs) occurred in ≥ 2 of 3 participants at a dose level, and/or ≥ 2 of 6 participants, at a dose level.
  Dose-limiting toxicity (DLT) was defined as a treatment-related (with possible, probable or definite attribution) Grade 3 to 5 CNS toxicity [Common Terminology Criteria for Adverse Events (CTCAE) v4] occurring within 30 days of stereotactic radiosurgery (SRS).
  The non-stratified outcome is reported as the number of DLTs observed in by radiation dose and by strata (Planning Target Volume (PTV) < 60 cm³ and from 60 to 150 cm³).
Time Frame: 30 days
Population: Participants receiving each radiotherapy level were stratified by tumor size.
Measure: Number; unit: Number of DLT observed
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 6 | 6 | 6 | 12
Number of DLT observed
  Planning Target Volume (PTV) < 60 cm³: number analyzed (Participants) | 3 | 3 | 3 | 6
  Planning Target Volume (PTV) < 60 cm³ | 0 | 0 | 0 | 1
  Planning Target Volume (PTV) 60 to 150 cm³: number analyzed (Participants) | 3 | 3 | 3 | 6
  Planning Target Volume (PTV) 60 to 150 cm³ | 0 | 0 | 0 | 1

2. Secondary Outcome: Number of Acute Toxicity Within 30 Days
Description: Acute toxicity is defined as treatment-related adverse events that occur within 30 days of receiving radiotherapy. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 is used to grade adverse events. The non-stratified outcome is reported as number of treatment-related adverse events observed for each radiotherapy dose level.
  Acute toxicity is based on radiotherapy dose level not tumor volume, and is reported by radiotherapy dose level only.
Time Frame: 30 days
Measure: Number; unit: adverse events
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 6 | 6 | 6 | 12
adverse events
  CTCAE Grade 1 | 5 | 2 | 2 | 4
  CTCAE Grade 2 | 0 | 0 | 1 | 0
  CTCAE Grade 3 | 0 | 0 | 1 | 0
  CTCAE Grade 4 | 0 | 0 | 0 | 1
  CTCAE Grade 5 | 0 | 0 | 0 | 1
  All grades | 5 | 2 | 4 | 6

3. Secondary Outcome: Long-term Toxicity After More Than 30 Days
Description: Long-term toxicity is defined as treatment-related adverse events (any grade or any Body System) that occur ≥ 30 days after receiving radiotherapy. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 is used to grade adverse events. The non-stratified outcome is reported as number of treatment-related adverse events observed for each dose level.
  Long-term toxicity is based on radiotherapy dose level not tumor volume, and is reported by radiotherapy dose level only.
Time Frame: 12 months
Measure: Number; unit: Number of adverse events
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 6 | 6 | 6 | 12
Number of adverse events
  CTCAE Grade 1 | 0 | 0 | 1 | 1
  CTCAE Grade 2 | 0 | 1 | 1 | 1
  CTCAE Grade 3 | 3 | 4 | 1 | 3
  CTCAE Grade 4 | 0 | 0 | 0 | 1
  All grades | 3 | 5 | 3 | 6

4. Secondary Outcome: Percent of Participants With Radiographic Response
Description: Radiographic response rate was assessed following radiotherapy until disease progression. Response is considered to be the sum and proportion participants that achieved a complete response (CR); partial response (PR); or minor response (MR). The outcome is expressed as a number without dispersion for each cohort.
  CR: Tumor is no longer detected by computed tomography (CT) or magnetic resonance imaging (MRI).
  PR: Decrease in the product of the two greatest diameters > 50%, as determined by CT or MRI, with no new lesions, and the same or lower dose of dexamethasone.
  MR: Decrease in the product of the two greatest diameters < 50%, as determined by CT or MRI, and neither PR nor PD.
  PD: New tumor lesion, or > 25% increase in the product of the two greatest diameters of target lesion, as determined by CT or MRI, provided that within 2 months of completion of radiotherapy, the participant has not had a decrease in steroid dose since the last evaluation.
Time Frame: 6 months
Measure: Number; unit: Percentage of participants
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 6 | 6 | 6 | 12
Percentage of participants
  Planning Target Volume (PTV) <60 CM3 | 100 | 100 | 100 | 33.3
  Planning Target Volume (PTV) 60-150CM3 | 66.7 | 66.7 | 66.7 | 16.7

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) following radiotherapy, measured in months. Progressive disease (PD) is defined as: New tumor lesion, or > 25% increase in the product of the 2 greatest diameters of target lesion, as determined by computed tomography (CT) or magnetic resonance imaging (MRI), provided that within 2 months of completion of radiotherapy, the participant has not had a decrease in steroid dose since the last evaluation. The outcome is expressed as the median with 95% confidence interval for each cohort.
Time Frame: 18 Months.
Population: Participants who have not progresses and have not reached reached 18 months post-treatment are not included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 3 | 3 | 3 | 6
Months
  Planning Target Volume (PTV) <60 CM3 | 13.4 [7.6 to 21.5] | 10.5 [8.7 to 11.7] | 33.5 [18.2 to 64.3] | 3.9 [1.7 to 21.2]
  Planning Target Volume (PTV) 60-150CM3 | 7.2 [3.2 to 23.3] | 6.5 [2.0 to 9.5] | 8.8 [5.6 to 17.6] | 4.0 [1.7 to 9.2]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed as those participants remaining alive with any tumor status following radiotherapy after 20 months. The outcome is stratified by Planning Target Volume (PTV) < 60 cm³ or 60 to 150 cm³, and expressed as the median value with 95% confidence interval.
Time Frame: 20 Months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 3 | 3 | 3 | 6
Months
  Planning Target Volume (PTV) <60 CM3 | 17.6 [14.9 to 27.8] | 19.9 [14.8 to 62.4] | 48.3 [33.5 to 64.4] | 10.2 [1.7 to 33]
  Planning Target Volume (PTV) 60-150CM3 | 10.1 [8.7 to 35.4] | 11.3 [10.9 to 16.1] | 17.6 [8.8 to 21.4] | 11.6 [5.3 to 12.7]

7. Secondary Outcome: Quality of Life by European Organisation for Research and Treatment of Cancer (EORTC-QLQ C30) Survey
Description: European Organization for Research and Treatment of Cancer (EORTC-QLQ C30) quality of life surveys were administered at study entry and 12 months after treatment initiation to assess health-related quality of life (HR-QOL). The EORTC-QLQ C30 survey has 30 questions and responses are on scale of 1 to 4 with 1 indicating "not at all" and 4 indicating "very much". The total score can range from 30 to 120. The outcome is stratified by Planning Target Volume (PTV) < 60 cm³ or 60 to 150 cm³, and is expressed as the mean of the difference from baseline to 12 months, with 95% confidence interval.
Time Frame: 12 Months
Population: Some participants did not contribute one or both of the baseline (study entry) and 12-month assessments, and the outcome (difference from baseline / study entry to 12 months after the start of treatment could not be calculated.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 5 | 6 | 6 | 11
score on a scale
  Planning Target Volume (PTV) <60 CM3: number analyzed (Participants) | 2 | 3 | 3 | 5
  Planning Target Volume (PTV) <60 CM3 | 41.6 [-275.9 to 359.3] | 58.3 [-16.3 to 132.9] | 80.5 [28.4 to 132.6] | 53.3 [14.2 to 92.4]
  Planning Target Volume (PTV) 60-150CM3: number analyzed (Participants) | 3 | 3 | 3 | 6
  Planning Target Volume (PTV) 60-150CM3 | 41.6 [-13.1 to 96.4] | 52.7 [0.68 to 104.8] | 44.4 [20.5 to 68.3] | 51.3 [13.7 to 89.07]

8. Secondary Outcome: Quality of Life by Brain-20 Survey
Description: Brain-20 (BN-20) quality of life surveys were administered at study entry and 12 months after treatment initiation to assess health-related quality of life (HR-QOL). The Brain-20 (BN-20) quality of life survey has 20 questions and responses are on scale of 1 to 4 with 1 indicating "not at all" (most favorable) and 4 indicating "very much" (least favorable). The total score can range from 20 to 80, and the result is expressed as the difference from baseline (study entry) to 12 months after the start of treatment. The outcome is stratified by Planning Target Volume (PTV) < 60 cm³ or 60 to 150 cm³, and expressed as the mean with 95% confidence interval.
Time Frame: 12 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 5 | 6 | 6 | 11
score on a scale
  Planning Target Volume (PTV) <60 CM3: number analyzed (Participants) | 2 | 3 | 3 | 5
  Planning Target Volume (PTV) <60 CM3 | 66.6 [-356.8 to 490.2] | 40.7 [-70.8 to 152.2] | 18.5 [-611.1 to 98.1] | 44.4 [-8.0 to 96.9]
  Planning Target Volume (PTV) 60-150CM3: number analyzed (Participants) | 3 | 3 | 3 | 6
  Planning Target Volume (PTV) 60-150CM3 | 40.7 [-1.4 to 82.9] | 55.5 [-43.9 to 155.0] | 59.2 [1.8 to 116.7] | 25.9 [-9.1 to 61.0]

9. Secondary Outcome: Quality of Life by MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) Survey
Description: MD Anderson Symptom Inventory - Brain Tumor (MDASI-BT) quality of life surveys were administered at study entry and 12 months after treatment initiation to assess health-related quality of life (HR-QOL). MDASI-BT quality of life survey has 23 questions and responses are on scale of 0 to 10 with 0 indicating "did not interfere" (most favorable) and 10 indicating "interfered completely" (least favorable). A participant's overall score is computed as the mean of that participant's individual scores, and can range 0 to 10. The outcome is stratified by Planning Target Volume (PTV) < 60 cm³ or 60 to 150 cm³, and expressed as the mean difference from baseline with 95% confidence interval. A positive value for the mean indicates worsening quality of life.
Time Frame: 12 months
Population: as for outcome 7
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 4 | 5 | 6 | 11
score on a scale
  Planning Target Volume (PTV) <60 CM3: number analyzed (Participants) | 2 | 2 | 3 | 5
  Planning Target Volume (PTV) <60 CM3 | 5.2 [-51.9 to 62.4] | 2.0 [-23.4 to 27.4] | 2.8 [-5.0 to 10.7] | 3.2 [0.2 to 6.3]
  Planning Target Volume (PTV) 60-150CM3: number analyzed (Participants) | 2 | 3 | 3 | 6
  Planning Target Volume (PTV) 60-150CM3 | 3.7 [0.5 to 6.9] | 3.2 [-5.1 to 11.6] | 2.3 [-3.0 to 7.6] | 3.6 [0.5 to 6.7]

10. Secondary Outcome: Treatment Failure Analysis
Description: Treatment failure in individual participants, ie, tumor recurrence or metastasis, can be described by the location relative to the first treatment failure (ie, infield, marginal, or distal), as further defined below.
  Failure pattern is defined as tumor recurrence or metastasis relative to the primary lesion that is
  * Infield: at tumor or within 5 mm
  * Marginal: > 5 mm or ≤ 20 mm from tumor
  * Distal: > 20 mm from tumor
  The outcome will be reported as the number of participants who failed treatment for each type of failure, ie, infield, marginal, or distal failure.
Time Frame: 18 months
Population: If the location of a participant's 1st treatment failure could not be determined, then a location assessment relative to any 2nd treatment failure can not done (null result), and for this reason, this analysis only includes participants for whom the location of the 1st treatment failure could be determined.
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
Number analyzed (Participants) | 6 | 6 | 4 | 11
Participants
  In-Field | 2 | 5 | 2 | 8
  Marginal | 1 | 0 | 1 | 1
  Distal | 3 | 1 | 1 | 2

ADVERSE EVENTS:
Arm/Group | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide
All-Cause Mortality (participants affected / at risk) | 6/6 | 5/6 | 4/6 | 10/12
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 0/6 | 9/12
Other Adverse Events (participants affected / at risk) | 6/6 | 5/6 | 6/6 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide (N=6) | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide (N=6) | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide (N=6) | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide (N=12)
Nervous system disorders-Other, altered mental state (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema cerebral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, ressection of recurrent tumor (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiosurgery (25 Gray x 5 Fractions)+Temozolomide (N=6) | Stereotactic Radiosurgery (30 Gray x 5 Fractions)+Temozolomide (N=6) | Stereotactic Radiosurgery (35 Gray x 5 Fractions)+Temozolomide (N=6) | Stereotactic Radiosurgery (40 Gray x 5 Fractions)+Temozolomide (N=12)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Nervous system disorders -Other, necrosis (Nervous system disorders) | 1 (1) | 1 (1) | 4 (4) | 2 (2)
Nervous system disorders -Other, aphasia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT01120639/Prot_SAP_000.pdf